CLINICAL TRIAL: NCT06887439
Title: Association of Endothelial Activation and Stress Index With Mortality and Poor Prognosis in Sepsis: A Prospective Observational Study
Brief Title: Association of EASIX in Sepsis
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mustafa Altınay, associate professor, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: iraz-24
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Sepsis; Septic Shock; Septic Syndrome
Keywords: sepsis; septic shock; endothelium
MeSH Terms: conditions — Sepsis; Shock, Septic; Toxemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sepsis group: Adult patients (≥18 years old) diagnosed with sepsis

SUMMARY:
This prospective study aims to determine the relationship between the EASIX score and mortality and prognosis in sepsis.

DETAILED DESCRIPTION:
Sepsis is a life-threatening condition characterized by a dysregulated host response to infection, leading to organ dysfunction. Despite advancements in medicine, sepsis remains a significant cause of death worldwide. An international study showed that 48.9 million sepsis cases were diagnosed in 195 countries between 1990 and 2017, resulting in 11 million deaths. Recent studies have demonstrated that early diagnosis and treatment reduce sepsis mortality. Therefore, research has focused on identifying biomarkers that aid in early diagnosis and prognosis.

The Endothelial Activation and Stress Index (EASIX) was first defined by Luft et al. as a biomarker reflecting endothelial damage. Calculated using readily available laboratory parameters-serum lactate dehydrogenase (LDH) level (U/L) x creatinine level (mg/dL) / platelet count (10⁹/L)-it has been commonly used to predict mortality and prognosis in hematological malignancies. Recently, its application in predicting sepsis mortality and prognosis has gained attention, although only limited retrospective studies have been published.

ELIGIBILITY:
Inclusion Criteria:

* • Patients diagnosed with sepsis during intensive care admission or admitted to intensive care with a diagnosis of sepsis

  * All patients over the age of 18

Exclusion Criteria:

* • Patients under the age of 18

  * Patients with a history of multiple intensive care admissions
  * Patients who died within 24 hours of diagnosis
  * Patients diagnosed with CRF or currently treated for ARF
  * Patients with deficient serum creatinine, LDH and platelet values at the time of diagnosis Patients for whom consent could not be obtained from themselves or their relatives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years old) diagnosed with sepsis were included.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
mortality | 28 days
  The primary finding of the study was 28-day mortality after sepsis diagnosis

SECONDARY OUTCOMES:
Septic shock | 28 days
  Septic shock was defined according to the SEPSIS-3 guidelines as the need for vasopressors or inotropes in patients diagnosed with sepsis.
Acute kidney injury | 28 days
  Acute kidney injury was defined according to KDIGO guidelines as a ≥0.3 mg/dL increase in serum creatinine over 48 hours, a ≥1.5-fold increase in serum creatinine over 7 days, or urine output <0.5 mL/kg/hour for 6 consecutive hours.

CONTACTS AND LOCATIONS:
Overall Officials: AYSE SURHAN CINAR, Study Chair — şişli etfal eğitim araştırma hastanesi
Locations (1):
- Sisli etfal research and training hospital, Istanbul, Turkey (Türkiye)